CLINICAL TRIAL: NCT00435214
Title: The HPV Persistence and Progression (PaP) Cohort at Kaiser Permanente Northern California
Brief Title: Human Papillomavirus (HPV) and Risk of Cervical Precancer and Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907079; 07-C-N079
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Cervical Neoplasia
Keywords: Cytology; papilloma virus; CIN; Screening; Cervix; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Discarded cervical Pap test specimens

SUMMARY:
Background:

* In most women, HPV infection does not cause symptoms and the infection goes away on its own. In a small percentage of women, the HPV infection does not go away and sometimes can result in cervical precancer or cancer.
* There are several different types of HPV. A better understanding of which types are related to cervical precancer and cancer may help guide doctors in clinical management of women who test positive for HPV and better understand why some women develop disease while others do not.

Objectives:

* To determine whether certain types of HPV are more risky than others and if so, whether they warrant separate detection in screening for cervical precancer and cancer.
* To determine if lasting infection by different HPV types carry different risk of cervical precancer and cancer.
* To determine what viral and genetic factors influence the development of cervical precancer and cancer.
* To evaluate new HPV tests and new biomarkers of cervical cancer risk.

Eligibility:

-Women 30 years of age and older who are in the cervical cancer screening program at the Kaiser Permanente health plan in Northern California. Women who tested positive for HPV and a random sample of women who tested negative for the virus are included.

Design:

-Data about participants genetic background and the type of carcinogenic HPV with which they are infected are analyzed.

DETAILED DESCRIPTION:
The carcinogenicity of the 15 HPV types with carcinogenic potential varies greatly. We wish to clarify clinical utility of carcinogenic HPV DNA testing in women 21 and older by understanding the unique properties of individual HPV genotypes for viral persistence and progression. Specifically, we seek to understand the timing and determinants of viral clearance versus persistence and, given persistence, the risk of progression to CIN3/cancer (greater than or equal to CIN3) among women infected with each type of carcinogenic HPV genotype at the ages when cancer occurs. The relevant natural history data are lacking. There are no NCI or other cohorts in which these and other questions are being adequately addressed.

Kaiser Permanente Northern California (KPNC) routinely uses a FDA-approved pooled-HPV genotype DNA test for carcinogenic HPV (Hybrid Capture 2 [HC2], Qiagen Corporation, Gaithersburg, MD) as an adjunct to cytology for cervical cancer screening in women 30 and older and as a triage for immediate colposcopy for women with equivocal Pap results at all ages. We are teaming with KPNC to create a carcinogenic HPV-positive cohort (HPV Persistence and Progression Cohort or PaP Cohort) for investigating the natural history of HPV genotypes. Specifically, we will store approximately 60,000 baseline specimens from the following sub-populations: 1) approximately 40,000 HPV positives and a random population sample of 4,000 baseline specimens from women aged 30 years and older; 2) approximately 5,000 HPV-orcytology-positives and random population sample of 2,000 baseline specimens from women aged 25-29 years of age; and 3) approximately 5,000 HPV-or cytology-positives and random population sample of 2,000 baseline specimens from women aged 21-24 years of age. We will use efficient sampling designs to achieve high power with minimal laboratory analyses, with specimens selected for testing based on clinical outcomes ascertained by linkage to the Kaiser cytology and histology databases and KPNC s active yearly follow-up of all HC2-positive women. We plan to "follow" women for three years after their enrollment in 2007-8 by banking their residual specimens collected at their return visits; longer follow-up would likely be biased by extensive censoring due to treatment.

Extremely low-cost specimen accrual, computerized follow-up using the KPNC databases, and leveraged funding will make this cohort highly cost-effective, with a proposed budget of $1,030,954 over 5 years. The de novo cost of screening this population to identify approximately 50,000 HPV-positive women 21 and older, which is performed by KPNC as part of routine screening and at no cost to us, is approximately $50 million. The clinical follow-up, cytology, and histologic diagnoses cost millions more. We can obtain genotyping and variant testing without cost to the Division of Cancer Epidemiology and Genetics (DCEG), via collaborations and the aforementioned Cooperative Agreement. The major costs are for personnel to save and handle the specimens, extraction of clinical and questionnaire data, and to offer women whose specimens have been banked an opt-out for use of the specimens.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women in KPNC aged 25 years or older who tested positive for HPV.

Will also include a random sample of women who tested negative for HPV.

EXCLUSION CRITERIA:

Male.

Children under 18.

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are teaming with Kaiser Permanente Northern California (KPNC) to create a carcinogenic HPV-positive cohort (HPV Persistence and Progression Cohort or PaP Cohort) for investigating the natural history of HPV genotypes. Specifically, we will store approximately 60,000 baseline specimens from the following sub-populations: 1) approximately 40,000 HPV positives and a random population sample of 4,000 baseline specimens from women aged 30 years and older; 2) approximately 5,000 HPV-or-cytologypositives and random population sample of 2,000 baseline specimens from women aged 25-29 years of age; and 3) approximately 5,000 HPV-or cytology-positives and random population sample of 2,000 baseline specimens from women aged 21-24 years of age.
Sampling Method: Probability Sample
Enrollment: 131110 (Actual)
Dates: Start 2007-01-29 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
CIN2+/CIN3+/Cancer | Ongoing
  Cervical histopathology; The detection of CIN2+,CIN3+, or cancer in histology results from tissue collected during cervical biopsies, excisional treatment or surgery.

SECONDARY OUTCOMES:
HPV Clearance | Ongoing
  HPV DNA testing:A negative HPV test result or normal cytology during follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Schiffman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

REFERENCES:
- [Background] Gage JC, Sadorra M, Lamere BJ, Kail R, Aldrich C, Kinney W, Fetterman B, Lorey T, Schiffman M, Castle PE; PaP Cohort Study Group. Comparison of the cobas Human Papillomavirus (HPV) test with the hybrid capture 2 and linear array HPV DNA tests. J Clin Microbiol. 2012 Jan;50(1):61-5. doi: 10.1128/JCM.05989-11. Epub 2011 Nov 9. PMID 22075592
- [Background] Wentzensen N, Sun C, Ghosh A, Kinney W, Mirabello L, Wacholder S, Shaber R, LaMere B, Clarke M, Lorincz AT, Castle PE, Schiffman M, Burk RD. Methylation of HPV18, HPV31, and HPV45 genomes and cervical intraepithelial neoplasia grade 3. J Natl Cancer Inst. 2012 Nov 21;104(22):1738-49. doi: 10.1093/jnci/djs425. Epub 2012 Oct 23. PMID 23093560
- [Background] Lamere BJ, Castle PE, Fetterman B, Poitras N, Stanley M, Shieh J, Lorey T, Kinney W, Schiffman M. A study of borderline positive Hybrid Capture 2 tests in the Kaiser Permanente Northern California cervical screening program: evidence against retesting. J Virol Methods. 2013 Apr;189(1):77-9. doi: 10.1016/j.jviromet.2013.01.011. Epub 2013 Feb 4. No abstract available. PMID 23384678